CLINICAL TRIAL: NCT02045966
Title: Effect of a Fixed Dose Combination Formulation of Daclatasvir/Asunaprevir/BMS-791325 on the Pharmacokinetics of a Cocktail of CYP Probe Substrates (Caffeine, Metoprolol, Montelukast, Flurbiprofen, Omeprazole, and Midazolam) and Transporter Probe Substrates (Digoxin and Pravastatin) in Healthy Subjects
Brief Title: Study to Determine the Potential DDIs When the Daclatasvir/Asunaprevir/BMS-791325 Three Drug Antiviral Combination Tablet (FDC) is Coadministered With a Cocktail of Cytochrome P450 (CYP) Probe Substrates and Transporter Probe Substrates (Digoxin and Pravastatin) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AI443-021
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: Cocktail + DCV 3DAA FDC + BMS-791325 (Experimental): Treatment A: Cocktail of CYP and transporter probe substrates orally as a single dose on Day 1
  Treatment B: DCV 3DAA FDC tablet administered orally BID on Days 6 to 15
  Treatment C: DCV 3DAA FDC tablet administered orally BID on Days 16 to 20, plus the cocktail of CYP and transporter probe substrates administered orally as a single dose on Day 16 only
  Treatment D: DCV 3DAA FDC tablet plus BMS-791325 75-mg single-agent tablet administered orally BID on Days 21 to 30
  Treatment E: DCV 3DAA FDC tablet plus BMS-791325 75-mg single-agent tablet administered orally BID on Days 31 to 35, plus the cocktail of CYP and transporter probe substrates administered orally as a single dose on Day 31 only
  Interventions: Drug: Cocktail; Drug: DCV 3DAA FDC; Drug: BMS-791325

INTERVENTIONS:
Drug: Cocktail — Cocktail = Caffeine 200 mg, Metoprolol 50 mg, Montelukast 10 mg, Flurbiprofen 50 mg, Omeprazole 40 mg, Midazolam 5 mg, Digoxin 0.25 mg, and Pravastatin 40 mg
Drug: DCV 3DAA FDC — DCV 30 mg + ASV 200 mg + BMS-791325 75 mg
Drug: BMS-791325

SUMMARY:
The primary purpose of this study is to assess the effect of the Daclatasvir/Asunaprevir/BMS-791325 fixed dose combination (FDC) tablet on the pharmacokinetics of the cocktail CYP and transporter probe substrates and to assess the effect of the DCV 3DAA FDC [DCV 3DAA FDC = fixed dose combination formulation of 3 direct-acting antivirals (3DAA) (DCV 30 mg, ASV 200 mg, and BMS-791325 75 mg)] + BMS-791325 75-mg single-agent tablet on the Pharmacokinetic (PK) of the cocktail CYP and transporter probe substrates.

DETAILED DESCRIPTION:
IND number: 79,599 and 101,943

Primary purpose: Other: study is being conducted to investigate the potential drug-drug interactions (DDIs) when the Daclatasvir/Asunaprevir/BMS-791325 FDC formulation is coadministered with a cocktail of cytochrome P450 (CYP) probe substrates (Caffeine, Metoprolol, Montelukast, Flurbiprofen, Omeprazole, and Midazolam) and transporter probe substrates (Digoxin and Pravastatin) in healthy subjects. It is also intended to characterize the PK of Daclatasvir (DCV), Asunaprevir (ASV), BMS-791325, and its major metabolite, BMS-794712, at steady state.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examinations, vital sign measurements, 12-lead ECG measurements, and clinical laboratory test results
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive. BMI = weight (kg)/[height (m)]2
* Men and women, ages 18 to 45 years, inclusive
* Women must not be of childbearing potential, must not be breastfeeding

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of important arrhythmias including, but not limited to, ventricular fibrillation, ventricular tachycardia, complete atrioventricular (A-V) block, Wolff-Parkinson-White syndrome
* History of cardiac arrhythmias or palpitations associated with presyncope or syncope, or history of unexplained syncope
* History of heart disease
* History of prolonged QT interval or torsades de pointes (TdP)
* History of hypokalemia
* Family history of sudden cardiac death at a young age, TdP, or Long QT syndrome
* History of asthma, bronchospasm, or sleep apnea
* History of rhabdomyolysis
* History of a bleeding disorder
* History of Raynaud's disease
* History of peptic ulcer disease or significant gastrointestinal bleed
* History of biliary disorders, including Gilbert's disease or Dubin-Johnson disease
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery (including cholecystectomy) that could impact upon the absorption of study drug

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] for each cocktail CYP and transporter probe substrate | 51 time points up to day 36

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) for each cocktail CYP and transporter probe substrate | 51 time points up to day 36
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] for each cocktail CYP and transporter probe substrate | 51 time points up to day 36
Cmax for the measured metabolites of the cocktail CYP and transporter probe substrates | 51 time points up to day 36
AUC(0-T) for the measured metabolites of the cocktail CYP and transporter probe substrates | 51 time points up to day 36
AUC(INF) for the measured metabolites of the cocktail CYP and transporter probe substrates | 51 time points up to day 36
Time of maximum observed concentration (Tmax) for each cocktail CYP and transporter probe substrate and their metabolites | 51 time points up to day 36
Half life (T-HALF) for each cocktail CYP and transporter probe substrate and their metabolites | 51 time points up to day 36
Ratio of metabolite Cmax to parent Cmax, corrected for molecular weight (MR_Cmax) for each cocktail CYP and transporter probe substrate and their metabolites | 51 time points up to day 36
Ratio of metabolite AUC(0-T) to parent AUC(0-T), corrected for molecular weight [MR_AUC(0-T)] for each cocktail CYP and transporter probe substrate and their metabolites | 51 time points up to day 36
Ratio of metabolite AUC(INF) to parent AUC(INF), corrected for molecular weight [MR_AUC(INF)] for each cocktail CYP and transporter probe substrate and their metabolites | 51 time points up to day 36
Apparent total body clearance (CLT/F) for each cocktail CYP and transporter probe substrate | 51 time points up to day 36
Cmax for Daclatasvir, Asunaprevir, BMS-791325, and the metabolite, BMS- 794712 at steady state | 24 time points up to day 31
Tmax for Daclatasvir, Asunaprevir, BMS-791325, and the metabolite, BMS- 794712 at steady state | 24 time points up to day 31
Concentration at 12 hours (C12) for Daclatasvir, Asunaprevir, BMS-791325, and the metabolite, BMS- 794712 at steady state | 24 time points up to day 31
Area under the concentration-time curve in one dosing interval [AUC(TAU)] for Daclatasvir, Asunaprevir, BMS-791325, and the metabolite, BMS- 794712 at steady state | 24 time points up to day 31
MR_Cmax for BMS-791325 and the metabolite, BMS-794712 | 24 time points up to day 31
Ratio of metabolite AUC(TAU) to parent AUC(TAU), corrected for molecular weight [MR_AUC(TAU)] for BMS-791325 and the metabolite, BMS-794712 | 24 time points up to day 31
Trough observed plasma concentration (Ctrough) for Daclatasvir, Asunaprevir, BMS-791325, and the metabolite, BMS-794712 | 24 time points up to day 31
Safety measured by the occurrence of AEs and SAEs, abnormalities in vital sign measurements exceeding pre-defined thresholds, findings on ECG measurements and physical examinations, and marked abnormalities in clinical laboratory test results | Up to day 36
  AEs = Adverse events
  SAEs = Serious Adverse events
  ECG = Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb